CLINICAL TRIAL: NCT00002611
Title: NATIONAL WILMS TUMOR STUDY-5 -- THERAPEUTIC TRIAL AND BIOLOGY STUDY
Brief Title: Combination Chemotherapy Alone or With Radiation Therapy in Treating Children With Kidney Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 9440; COG-Q9401 (Other: Children's Oncology Group); NWTS-Q9401 (Other: NWTS); CCG-4941 (Other: Children's Cancer Group); POG-9440 (Other: Pediatric Oncology Group); INT-0150; NWTS-5 (Other: NWTS); CDR0000063901 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2014-07

CONDITIONS: Kidney Cancer
Keywords: stage I Wilms tumor; stage II Wilms tumor; stage III Wilms tumor; stage IV Wilms tumor; stage V Wilms tumor; clear cell sarcoma of the kidney
MeSH Terms: conditions — Kidney Neoplasms; Wilms Tumor | interventions — Dactinomycin; Filgrastim; Cyclophosphamide; Doxorubicin; Etoposide; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Stratum 1 (Active Comparator): Stage I favorable histology (FH) Wilms' tumor, under 24 months of age, and tumor weight less than 550 g: After conventional surgery (nephrectomy), patients receive regimen EE-4A comprising dactinomycin (DACT) IV weekly on weeks 0, 3, 6, 9, 12, 15, and 18 and vincristine sulfate (VCR) IV weekly on weeks 1-10, 12, 15, and 18.
  Interventions: Biological: dactinomycin; Drug: vincristine sulfate; Procedure: conventional surgery
- Stratum 2 (Active Comparator): Stage I FH Wilms' tumor and age 24 months and over or tumor weight at least 550 g; stage I focal anaplastic (FA) or diffuse anaplastic (DA) Wilms' tumor: Patients receive regimen EE-4A comprising dactinomycin (DACT) IV weekly on weeks 0, 3, 6, 9, 12, 15, and 18 and vincristine sulfate (VCR) IV weekly on weeks 1-10, 12, 15, and 18.
  Interventions: Biological: dactinomycin; Drug: vincristine sulfate
- Stratum 3 (Active Comparator): Stage II FH Wilms' tumor: Patients receive regimen EE-4A comprising dactinomycin (DACT) IV weekly on weeks 0, 3, 6, 9, 12, 15, and 18 and vincristine sulfate (VCR) IV weekly on weeks 1-10, 12, 15, and 18.
  Interventions: Biological: dactinomycin; Drug: vincristine sulfate
- Stratum 4 (Active Comparator): Stage III FH Wilms' tumor; stage II or III FA Wilms' tumor: After conventional surgery (nephrectomy), patients receive regimen DD-4A comprising dactinomycin DACT IV weekly on weeks 0, 6, 12, 18, and 24; doxorubicin hydrochloride IV weekly on weeks 3, 9, 15, and 21; and vincristine sulfate VCR IV weekly on weeks 1-10, 12, 15, 18, 21, and 24. Patients also undergo abdominal radiation therapy.
  Interventions: Biological: dactinomycin; Drug: doxorubicin hydrochloride; Drug: vincristine sulfate; Procedure: conventional surgery; Radiation: radiation therapy
- Stratum 5 (Active Comparator): Stage IV FH or FA Wilms' tumor: patients receive regimen DD-4A comprising dactinomycin DACT IV weekly on weeks 0, 6, 12, 18, and 24; doxorubicin hydrochloride IV weekly on weeks 3, 9, 15, and 21; and vincristine sulfate VCR IV weekly on weeks 1-10, 12, 15, 18, 21, and 24. Patients also undergo abdominal radiation therapy, and whole lung radiation therapy (at the discretion of the investigator).
  Interventions: Biological: dactinomycin; Drug: doxorubicin hydrochloride; Drug: vincristine sulfate
- Stratum 6 (Active Comparator): Stage V FH, FA, or DA Wilms' tumor: After bilateral conventional surgery (biopsy), patients with FH receive chemotherapy as in stratum 1 (dactinomycin IV weeks 0, 3, 6, 9, 12, 15, and 18 and vincristine sulfate IV weeks 1-10, 12, 15, and 18) or 4 (dactinomycin IV weeks 0, 6, 12, 18, and 24; doxorubicin hydrochloride IV weeks 3, 9, 15, and 21; and vincristine sulfate VCR IV weeks 1-10, 12, 15, 18, 21, and 24). Patients with FA or DA receive chemotherapy as in stratum 7 (vincristine sulfate VCR IV weeks 1, 2, 4-8, 10-13, 18, and 24; cyclophosphamide sulfate (CTX) IV over 1 hour on days 1-3 of weeks 6, 12, 18, and 24 and on days 1-5 of weeks 3, 9, 15, and 21; doxorubicin hydrochloride IV (beginning after CTX infusion) weeks 0, 6, 12, 18, and 24; and etoposide (VP-16) IV over 1 hour (beginning after CTX infusion) on days 1-5 of weeks 3, 9, 15, and 21. Filgrastim (G-CSF) is administered subcutaneously (SC) beginning 24 hours after completion of chemotherapy.
  Interventions: Biological: dactinomycin; Biological: filgrastim; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: vincristine sulfate; Procedure: conventional surgery
- Stratum 7 (Active Comparator): Stages I-IV clear cell sarcoma): After conventional surgery (nephrectomy), patients receive vincristine sulfate VCR IV weekly on weeks 1, 2, 4-8, 10-13, 18, and 24; cyclophosphamide sulfate (CTX) IV over 1 hour on days 1-3 of weeks 6, 12, 18, and 24 and on days 1-5 of weeks 3, 9, 15, and 21; doxorubicin hydrochloride IV (beginning after CTX infusion) weekly on weeks 0, 6, 12, 18, and 24; and etoposide (VP-16) IV over 1 hour (beginning after CTX infusion) on days 1-5 of weeks 3, 9, 15, and 21. Filgrastim (G-CSF) is administered subcutaneously (SC) beginning 24 hours after completion of chemotherapy and continuing until blood counts recover. Patients also undergo abdominal radiotherapy and whole lung radiotherapy (if pulmonary metastases are present).
  Interventions: Biological: filgrastim; Drug: doxorubicin hydrochloride; Drug: etoposide; Procedure: conventional surgery; Radiation: radiation therapy
- Stratum 8 (Active Comparator): Stages II-IV DA Wilms' tumor: After conventional surgery (nephrectomy), Patients receive treatment as in stratum 7 (patients receive vincristine sulfate VCR IV weekly on weeks 1, 2, 4-8, 10-13, 18, and 24; cyclophosphamide sulfate (CTX) IV over 1 hour on days 1-3 of weeks 6, 12, 18, and 24 and on days 1-5 of weeks 3, 9, 15, and 21; doxorubicin hydrochloride IV (beginning after CTX infusion) weekly on weeks 0, 6, 12, 18, and 24; and etoposide (VP-16) IV over 1 hour (beginning after CTX infusion) on days 1-5 of weeks 3, 9, 15, and 21. Filgrastim (G-CSF) is administered subcutaneously (SC) beginning 24 hours after completion of chemotherapy and continuing until blood counts recover. Patients also undergo abdominal radiotherapy and whole lung radiotherapy (if pulmonary metastases are present).
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: vincristine sulfate; Procedure: conventional surgery; Radiation: radiation therapy
- Stratum 9 (Active Comparator): Stages I-IV rhabdoid tumor: After conventional surgery (nephrectomy), patients receive carboplatin IV on days 1-2 and VP-16 IV over 1 hour (beginning after carboplatin infusion) on days 1-3 of weeks 0, 3, 9, 12, 18, and 21 and CTX IV over 1 hour on days 1-5 of weeks 6, 15, and 24. Filgrastim G-CSF is administered as on stratum 7. Patients also undergo radiation therapy. After completion of chemotherapy, patients undergo second-look conventional surgery (laparotomy) and conventional surgery (partial nephrectomy or wedge excision if feasible). After conventional surgery (second-look surgery), patients without persistent or residual disease resume chemotherapy.
  Interventions: Biological: filgrastim; Drug: etoposide; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Biological: dactinomycin
  Arms: Stratum 1; Stratum 2; Stratum 3; Stratum 4; Stratum 5; Stratum 6
Biological: filgrastim
  Arms: Stratum 6; Stratum 7; Stratum 8; Stratum 9
Drug: cyclophosphamide
  Arms: Stratum 6; Stratum 8
Drug: doxorubicin hydrochloride — Source and Pharmacology: An anthracycline antibiotic isolated from cultures of Streptomyces peucetius. Binds to DNA and inhibits nucleic acid synthesis, with its major lethal effect occurring during the S phase of the cell cycle. Has some topoisomerase II inhibitory activity. Since it is primarily excreted by the liver, any liver impairment may enhance toxicity. 40% to 50% is excreted in the bile; <5% in the urine. The drug has a very short initial t½ of <20 minutes and a terminal t½ of 17 hours. Animal studies indicate cytotoxic levels persist in tissue for as long as 24 hours.
  Other Names: NSC #123127; (Adriamycin)
  Arms: Stratum 4; Stratum 5; Stratum 6; Stratum 7; Stratum 8
Drug: etoposide
  Arms: Stratum 6; Stratum 7; Stratum 8; Stratum 9
Drug: vincristine sulfate
  Arms: Stratum 1; Stratum 2; Stratum 3; Stratum 4; Stratum 5; Stratum 6; Stratum 8
Procedure: conventional surgery
  Arms: Stratum 1; Stratum 4; Stratum 6; Stratum 7; Stratum 8; Stratum 9
Radiation: radiation therapy
  Arms: Stratum 4; Stratum 7; Stratum 8; Stratum 9

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high energy x-rays to damage tumor cells. It is not yet known whether combination chemotherapy alone or combination chemotherapy plus radiation therapy is more effective for childhood kidney cancer.

PURPOSE: Phase III trial to compare the effectiveness of combination chemotherapy with or without radiation therapy in treating children who have kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Increase survival rate of children with favorable histology (FH) Wilms' tumor and other childhood renal tumors.
* Determine whether loss of heterozygosity for chromosome 16q or 1p in tumor tissue is associated with a poorer prognosis in children with FH Wilms' tumor.
* Determine whether increased DNA content in tumor cells is associated with a poorer prognosis in children with FH Wilms' tumor.
* Decrease the acute and long-term morbidity in children with Wilms' tumor by limiting initial therapy and consistently using the same regimen (protocol NWTS-5/R) for patients who relapse following initial treatment.
* Improve overall and disease-free survival of patients with renal tumors of unfavorable histology, including Wilms' tumor with diffuse anaplasia and clear cell sarcoma of the kidney, using a new treatment regimen that includes etoposide (VP-16) and cyclophosphamide (CTX).
* Improve overall and disease-free survival in patients with malignant rhabdoid tumor of the kidney using a new treatment regimen that includes carboplatin, VP-16, and CTX. (The rhabdoid tumor stratum closed to accrual effective 07/13/2001)
* Provide data regarding loss of heterozygosity for chromosomes 11p15, 16q, and 1p, age at diagnosis, precursor lesions (perilobar, intralobar, nephroblastomatosis), bilaterality, and presence of congenital anomalies required for the completion of protocol A0026 (a case-control study of risk factors for Wilms' tumor).

OUTLINE: This is a multicenter study. Patients are assigned to one of nine strata based on tumor histology, stage, tumor weight, and age.

* Stratum 1 (stage I favorable histology (FH) Wilms' tumor, under 24 months of age, and tumor weight less than 550 g): After nephrectomy, patients receive regimen EE-4A comprising dactinomycin (DACT) IV weekly on weeks 0, 3, 6, 9, 12, 15, and 18 and vincristine (VCR) IV weekly on weeks 1-10, 12, 15, and 18.
* Stratum 2 (stage I FH Wilms' tumor and age 24 months and over or tumor weight at least 550 g; stage I focal anaplastic (FA) or diffuse anaplastic (DA) Wilms' tumor): Patients receive therapy as in stratum 1.
* Stratum 3 (stage II FH Wilms' tumor): Patients receive therapy as in stratum 1.
* Stratum 4 (stage III FH Wilms' tumor; stage II or III FA Wilms' tumor): After nephrectomy, patients receive regimen DD-4A comprising DACT IV weekly on weeks 0, 6, 12, 18, and 24; doxorubicin IV weekly on weeks 3, 9, 15, and 21; and VCR IV weekly on weeks 1-10, 12, 15, 18, 21, and 24. Patients also undergo abdominal radiotherapy.
* Stratum 5 (stage IV FH or FA Wilms' tumor): Patients receive chemotherapy as in stratum 4, abdominal radiotherapy, and whole lung radiotherapy (at the discretion of the investigator).
* Stratum 6 (stage V FH, FA, or DA Wilms' tumor ): After bilateral biopsy, patients with FH receive chemotherapy as in stratum 1 or 4. Patients with FA or DA receive chemotherapy as in stratum 7.
* Stratum 7 (stages I-IV clear cell sarcoma): After nephrectomy, patients receive VCR IV weekly on weeks 1, 2, 4-8, 10-13, 18, and 24; cyclophosphamide (CTX) IV over 1 hour on days 1-3 of weeks 6, 12, 18, and 24 and on days 1-5 of weeks 3, 9, 15, and 21; doxorubicin IV (beginning after CTX infusion) weekly on weeks 0, 6, 12, 18, and 24; and etoposide (VP-16) IV over 1 hour (beginning after CTX infusion) on days 1-5 of weeks 3, 9, 15, and 21. Filgrastim (G-CSF) is administered subcutaneously (SC) beginning 24 hours after completion of chemotherapy and continuing until blood counts recover. Patients also undergo abdominal radiotherapy and whole lung radiotherapy (if pulmonary metastases are present).
* Stratum 8 (stages II-IV DA Wilms' tumor): Patients receive treatment as in stratum 7.
* Stratum 9 (stages I-IV rhabdoid tumor): After nephrectomy, patients receive carboplatin IV on days 1-2 and VP-16 IV over 1 hour (beginning after carboplatin infusion) on days 1-3 of weeks 0, 3, 9, 12, 18, and 21 and CTX IV over 1 hour on days 1-5 of weeks 6, 15, and 24. G-CSF is administered as in stratum 7. Patients also undergo radiotherapy. (The rhabdoid tumor stratum closed to accrual effective 07/13/2001.) After completion of chemotherapy, patients undergo second-look laparotomy and partial nephrectomy or wedge excision (if feasible). After second-look surgery, patients without persistent or residual disease resume chemotherapy.

Patients are followed every 3 months for 5 years, every 6 months for 2 years, and then annually for 3 years.

PROJECTED ACCRUAL: A total of 207 patients will be accrued for the treatment portion of this study. (The rhabdoid tumor stratum closed to accrual effective 07/13/2001.)

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage I-V kidney cancer of one of the following histologies:

  * Wilms' tumor, favorable histology
  * Wilms' tumor, focal or diffuse anaplastic
  * Clear cell sarcoma
  * Rhabdoid tumor

    * (The rhabdoid tumor stratum closed to accrual effective 07/13/2001)
* Prior nephrectomy or biopsy required

  * Prior bilateral biopsy (preferably open) with bilateral staging and pathologic evaluation required for bilateral tumor
* Must begin study therapy within 5 days after nephrectomy (unless medically contraindicated)

PATIENT CHARACTERISTICS:

Age:

* Under 16

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* See Disease Characteristics

Ages: 0 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3031 (Actual)
Dates: Start 1995-07; Primary Completion 2002-06 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M. Green, MD, Study Chair — Roswell Park Cancer Institute
Locations (235):
- United States (206):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - University of South Alabama Medical Center, Mobile, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital of Oakland, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center/Kaiser Foundation Hospital - San Diego, San Diego, California
  - Children's Hospital San Diego, San Diego, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Children's Hospital of Denver, Denver, Colorado
  - Childhood Hematology/Oncology Associates, Denver, Colorado
  - Presbyterian-St Luke's Medical Center, Denver, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Alfred I. Dupont Institute, Wilmington, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - Joe DiMaggio Children's Hospital at Memorial, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami-Jackson Memorial Hospital, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Nemours Children's Clinic-Orlando, Orlando, Florida
  - Sacred Heart Children's Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Tampa Children's Hospital, Tampa, Florida
  - St. Mary's Hospital, West Palm Beach, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Children's Healthcare of Atlanta - Scottish Rite, Atlanta, Georgia
  - Medical College of Georgia Comprehensive Cancer Center, Augusta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Memorial Health University Medical Center, Inc., Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Mountain States Tumor Institute, Boise, Idaho
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Hope Children's Hospital, Oak Lawn, Illinois
  - Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - St. Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Raymond Blank Memorial Hospital for Children, Des Moines, Iowa
  - John Stoddard Cancer Center, Des Moines, Iowa
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Wesley Medical Center, Wichita, Kansas
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Ochsner Clinic, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health and DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Mary's/Duluth Clinic Cancer Center, Duluth, Minnesota
  - Children's Hospitals and Clinics - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Hospitals and Clinics of Minnesota, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Atlantic Health System, Summit, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - State University of New York Health Science Center at Brooklyn College of Medicine, Brooklyn, New York
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia Presbyterian Hospital, New York, New York
  - James P. Wilmot Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Saint Joseph's Health System, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Dakota Cancer Institute, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Forum Health-Tod Childrens Hospital, Youngstown, Ohio
  - Children's Hospital of Oklahoma, Oklahoma City, Oklahoma
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - Doernbecher Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sioux Valley Hospital, Sioux Falls, South Dakota
  - East Tennessee State University Cancer Center at JCMC, Johnson City, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Children's Hospital of Austin, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Health Care System, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Vermont Cancer Center, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Carilion Medical Center for Children, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Cooperative, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Mary Bridge Children's Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University - Charleston, Charleston, West Virginia
  - Cabell-Huntington Hospital, Inc, Huntington, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (6):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (16):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Laval University Medical Center, Sainte-Foy, Quebec
  - Centre Hospitalier de L'Universite Laval, Sainte-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- Starship Children's Hospital, Auckland, New Zealand
- Puerto Rico (2):
  - University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan
  - San Jorge Childrens Hospital, Santurce
- Switzerland (3):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva
  - Swiss Pediatric Oncology Group Lausanne, Lausanne

REFERENCES:
- [Background] Grundy PE, Green DM, Dirks AC, Berendt AE, Breslow NE, Anderson JR, Dome JS. Clinical significance of pulmonary nodules detected by CT and Not CXR in patients treated for favorable histology Wilms tumor on national Wilms tumor studies-4 and -5: a report from the Children's Oncology Group. Pediatr Blood Cancer. 2012 Oct;59(4):631-5. doi: 10.1002/pbc.24123. Epub 2012 Mar 15. PMID 22422736
- [Background] Kieran K, Anderson JR, Dome JS, Ehrlich PF, Ritchey ML, Shamberger RC, Perlman EJ, Green DM, Davidoff AM. Lymph node involvement in Wilms tumor: results from National Wilms Tumor Studies 4 and 5. J Pediatr Surg. 2012 Apr;47(4):700-6. doi: 10.1016/j.jpedsurg.2011.08.017. PMID 22498384
- [Background] Lange J, Peterson SM, Takashima JR, Grigoriev Y, Ritchey ML, Shamberger RC, Beckwith JB, Perlman E, Green DM, Breslow NE. Risk factors for end stage renal disease in non-WT1-syndromic Wilms tumor. J Urol. 2011 Aug;186(2):378-86. doi: 10.1016/j.juro.2011.03.110. Epub 2011 Jun 17. PMID 21683387
- [Background] Kalapurakal JA, Green DM, Haase G, Anderson JR, Dome JS, Grundy PE. Outcomes of children with favorable histology wilms tumor and peritoneal implants treated in National Wilms Tumor Studies-4 and -5. Int J Radiat Oncol Biol Phys. 2010 Jun 1;77(2):554-8. doi: 10.1016/j.ijrobp.2009.04.081. PMID 20457352
- [Background] Ehrlich PF, Ferrer FA, Ritchey ML, Anderson JR, Green DM, Grundy PE, Dome JS, Kalapurakal JA, Perlman EJ, Shamberger RC. Hepatic metastasis at diagnosis in patients with Wilms tumor is not an independent adverse prognostic factor for stage IV Wilms tumor: a report from the Children's Oncology Group/National Wilms Tumor Study Group. Ann Surg. 2009 Oct;250(4):642-8. doi: 10.1097/SLA.0b013e3181b76f20. PMID 19730241
- [Background] Ritchey M, Daley S, Shamberger RC, Ehrlich P, Hamilton T, Haase G, Sawin R; National Wilms' Tumor Study Group. Ureteral extension in Wilms' tumor: a report from the National Wilms' Tumor Study Group (NWTSG). J Pediatr Surg. 2008 Sep;43(9):1625-9. doi: 10.1016/j.jpedsurg.2008.01.067. PMID 18778996
- [Background] van den Heuvel-Eibrink MM, Grundy P, Graf N, Pritchard-Jones K, Bergeron C, Patte C, van Tinteren H, Rey A, Langford C, Anderson JR, de Kraker J. Characteristics and survival of 750 children diagnosed with a renal tumor in the first seven months of life: A collaborative study by the SIOP/GPOH/SFOP, NWTSG, and UKCCSG Wilms tumor study groups. Pediatr Blood Cancer. 2008 Jun;50(6):1130-4. doi: 10.1002/pbc.21389. PMID 18095319
- [Background] Breslow NE, Beckwith JB, Perlman EJ, Reeve AE. Age distributions, birth weights, nephrogenic rests, and heterogeneity in the pathogenesis of Wilms tumor. Pediatr Blood Cancer. 2006 Sep;47(3):260-7. doi: 10.1002/pbc.20891. PMID 16700047
- [Background] Kalapurakal JA, Nan B, Norkool P, Coppes M, Perlman E, Beckwith B, Ritchey M, Breslow N, Grundy P, D'angio GJ, Green DM, Thomas PR. Treatment outcomes in adults with favorable histologic type Wilms tumor-an update from the National Wilms Tumor Study Group. Int J Radiat Oncol Biol Phys. 2004 Dec 1;60(5):1379-84. doi: 10.1016/j.ijrobp.2004.05.057. PMID 15590168
- [Result] Gadd S, Huff V, Huang CC, Ruteshouser EC, Dome JS, Grundy PE, Breslow N, Jennings L, Green DM, Beckwith JB, Perlman EJ. Clinically relevant subsets identified by gene expression patterns support a revised ontogenic model of Wilms tumor: a Children's Oncology Group Study. Neoplasia. 2012 Aug;14(8):742-56. doi: 10.1593/neo.12714. PMID 22952427
- [Result] Perlman EJ, Grundy PE, Anderson JR, Jennings LJ, Green DM, Dome JS, Shamberger RC, Ruteshouser EC, Huff V. WT1 mutation and 11P15 loss of heterozygosity predict relapse in very low-risk wilms tumors treated with surgery alone: a children's oncology group study. J Clin Oncol. 2011 Feb 20;29(6):698-703. doi: 10.1200/JCO.2010.31.5192. Epub 2010 Dec 28. PMID 21189373
- [Result] Fernandez CV, Anderson J, Breslow NE, Dome JS, Grundy PE, Perlman EJ, Green DM; National Wilms Tumor Study Group/Children's Oncology Group. Anthropomorphic measurements and event-free survival in patients with favorable histology Wilms tumor: a report from the Children's Oncology Group. Pediatr Blood Cancer. 2009 Feb;52(2):254-8. doi: 10.1002/pbc.21809. PMID 18989885
- [Result] Huang CC, Gadd S, Breslow N, Cutcliffe C, Sredni ST, Helenowski IB, Dome JS, Grundy PE, Green DM, Fritsch MK, Perlman EJ. Predicting relapse in favorable histology Wilms tumor using gene expression analysis: a report from the Renal Tumor Committee of the Children's Oncology Group. Clin Cancer Res. 2009 Mar 1;15(5):1770-8. doi: 10.1158/1078-0432.CCR-08-1030. Epub 2009 Feb 10. PMID 19208794
- [Result] Malogolowkin M, Cotton CA, Green DM, Breslow NE, Perlman E, Miser J, Ritchey ML, Thomas PR, Grundy PE, D'Angio GJ, Beckwith JB, Shamberger RC, Haase GM, Donaldson M, Weetman R, Coppes MJ, Shearer P, Coccia P, Kletzel M, Macklis R, Tomlinson G, Huff V, Newbury R, Weeks D; National Wilms Tumor Study Group. Treatment of Wilms tumor relapsing after initial treatment with vincristine, actinomycin D, and doxorubicin. A report from the National Wilms Tumor Study Group. Pediatr Blood Cancer. 2008 Feb;50(2):236-41. doi: 10.1002/pbc.21267. PMID 17539021
- [Result] Dome JS, Cotton CA, Perlman EJ, Breslow NE, Kalapurakal JA, Ritchey ML, Grundy PE, Malogolowkin M, Beckwith JB, Shamberger RC, Haase GM, Coppes MJ, Coccia P, Kletzel M, Weetman RM, Donaldson M, Macklis RM, Green DM. Treatment of anaplastic histology Wilms' tumor: results from the fifth National Wilms' Tumor Study. J Clin Oncol. 2006 May 20;24(15):2352-8. doi: 10.1200/JCO.2005.04.7852. PMID 16710034
- [Result] Ehrlich PF, Hamilton TE, Grundy P, Ritchey M, Haase G, Shamberger RC; National Wilms' Tumor Study Group (National Wilms' Tumor Study 5). The value of surgery in directing therapy for patients with Wilms' tumor with pulmonary disease. A report from the National Wilms' Tumor Study Group (National Wilms' Tumor Study 5). J Pediatr Surg. 2006 Jan;41(1):162-7; discussion 162-7. doi: 10.1016/j.jpedsurg.2005.10.020. PMID 16410127
- [Result] Seibel NL, Sun J, Anderson JR, et al.: Outcome of clear cell sarcoma of the kidney (CCSK) treated on the National Wilms Tumor Study-5 (NWTS). [Abstract] J Clin Oncol 24 (Suppl 18): A-9000, 502s, 2006.
- [Result] Dome JS, Bockhold CA, Li SM, Baker SD, Green DM, Perlman EJ, Hill DA, Breslow NE. High telomerase RNA expression level is an adverse prognostic factor for favorable-histology Wilms' tumor. J Clin Oncol. 2005 Dec 20;23(36):9138-45. doi: 10.1200/JCO.2005.00.562. Epub 2005 Sep 19. PMID 16172460
- [Result] Ehrlich PF, Ritchey ML, Hamilton TE, Haase GM, Ou S, Breslow N, Grundy P, Green D, Norkool P, Becker J, Shamberger RC. Quality assessment for Wilms' tumor: a report from the National Wilms' Tumor Study-5. J Pediatr Surg. 2005 Jan;40(1):208-12; discussion 212-3. doi: 10.1016/j.jpedsurg.2004.09.044. PMID 15868587
- [Result] Grundy PE, Breslow NE, Li S, Perlman E, Beckwith JB, Ritchey ML, Shamberger RC, Haase GM, D'Angio GJ, Donaldson M, Coppes MJ, Malogolowkin M, Shearer P, Thomas PR, Macklis R, Tomlinson G, Huff V, Green DM; National Wilms Tumor Study Group. Loss of heterozygosity for chromosomes 1p and 16q is an adverse prognostic factor in favorable-histology Wilms tumor: a report from the National Wilms Tumor Study Group. J Clin Oncol. 2005 Oct 10;23(29):7312-21. doi: 10.1200/JCO.2005.01.2799. Epub 2005 Aug 29. PMID 16129848
- [Result] Miller MA, Karacay B, Breslow NE, Li S, O'Dorisio MS, Grundy PE, Sandler AD. Prognostic value of quantifying apoptosis factor expression in favorable histology wilms tumors. J Pediatr Hematol Oncol. 2005 Jan;27(1):11-4. doi: 10.1097/01.mph.0000149961.71266.27. PMID 15654272
- [Derived] Benedetti DJ, Varela CR, Renfro LA, Tornwall B, Dix DB, Ehrlich PF, Glick RD, Kalapurakal J, Perlman E, Gratias E, Seibel NL, Geller JI, Khanna G, Malogolowkin M, Grundy P, Fernandez CV, Dome JS, Mullen EA. Treatment of children with favorable histology Wilms tumor with extrapulmonary metastases: A report from the COG studies AREN0533 and AREN03B2 and NWTSG study NWTS-5. Cancer. 2024 Mar 15;130(6):947-961. doi: 10.1002/cncr.35099. Epub 2023 Nov 7. PMID 37933882
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/